CLINICAL TRIAL: NCT01911728
Title: A Phase I Open-label Study to Evaluate the Effect of Multiple Doses of MDV3100 (ASP9785) on the Pharmacokinetics of Substrates for CYP2C8, CYP2C9, CYP2C19, and CYP3A4 in Patients With Castration-resistant Prostate Cancer
Brief Title: Drug-drug Interaction Study With MDV3100 and a Cocktail of Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0007; 2011-000163-26 (EudraCT Number)
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Pharmacokinetics of MDV3100; Castration Resistant Prostate Cancer (CRPC)
Keywords: Drug-Drug Interaction; Phase 1; MDV3100; Xtandi; Enzalutamide
MeSH Terms: interventions — enzalutamide; Pioglitazone; Warfarin; Omeprazole; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multiple doses of MDV3100 (Experimental): Multiple doses of MDV3100 and a single dose of pioglitazone and a single dose of cocktail containing -warfarin, omeprazole and midazolam
  Interventions: Drug: MDV3100; Drug: Pioglitazone; Drug: Warfarin; Drug: Omeprazole; Drug: Midazolam

INTERVENTIONS:
Drug: MDV3100 — Oral
  Other Names: Xtandi; enzalutamide
Drug: Pioglitazone — Oral
Drug: Warfarin — Oral
Drug: Omeprazole — Oral
Drug: Midazolam — Oral

SUMMARY:
A drug-drug interaction study to investigate the potential pharmacokinetic interaction between MDV3100 and a cocktail of substrates for pioglitazone (CYP2C8 substrate), S-warfarin (CYP2C9 substrate), omeprazole (CYP2C19 substrate), and midazolam (CYP3A4 substrate).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features;
* Ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., medical or surgical castration);
* Progressive disease by prostate specific antigen (PSA) or imaging whether or not after chemotherapy in the setting of medical or surgical castration. Disease progression for study entry is defined as one or more of the following 3 criteria:

  * PSA progression defined by a minimum of 3 rising PSA levels with an interval of ≥1 week between each determination. The PSA value during the pre investigational period should be ≥2 μg/L (2 ng/mL);
  * Soft tissue disease progression defined by the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) for soft tissue disease (see Appendix A);
  * Bone disease progression defined by two or more new lesions on bone scan.

Exclusion Criteria:

* Confirmed CYP2C8, CYP2C9, or CYP2C19 poor metabolizer status based on genotyping analysis;
* Absolute neutrophil count < 1,500/μL, platelet count < 100,000/μL, and hemoglobin < 5.6 mmol/L (9 g/dL) during the screening period (NOTE: patients may not have received any growth factors or blood transfusions within 7 days prior to the hematologic laboratory values obtained during the screening period);
* Total bilirubin > 1.5 times, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal during the screening period;
* Creatinine > 177 μmol/L (2 mg/dL) during the screening period;
* Albumin < 30 g/L (3.0 g/dL) during the screening period;
* Treatment with androgen receptor antagonists (bicalutamide, flutamide, nilutamide), 5 α reductase inhibitors (finasteride, dutasteride), estrogens, or chemotherapy within 4 weeks prior to enrollment (Day 1 visit) or plans to initiate treatment with any of these treatments during the study;
* Use of herbal products that may decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone/prednisolone per day within 4 weeks prior to enrollment (Day 1 visit) or plans to initiate treatment with any of these treatments during the study;
* Structurally unstable bone lesions suggesting impending fracture;
* History of seizure, including any febrile seizure, loss of consciousness, or transient ischemia attack within 12 months prior to enrollment (Day 1 visit), or any condition that may pre-dispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-07-25 (Actual); Primary Completion 2012-02-21 (Actual); Study Completion 2012-02-21 (Actual)

PRIMARY OUTCOMES:
Assessment of the pharmacokinetic profile of pioglitazone (CYP2C8 substrate) in combination with MDV3100 PTM and MDV3100 | Day 1 through Day 72 (75 times)
  (Maximum concentration (observed))Cmax, (Area Under Curve from the time of dosing to the last measurable concentration)AUC0-t, (AUC extrapolated to infinity)AUC0-inf
Assessment of the pharmacokinetic profile of S-warfarin (CYP2C9 substrate) in combination with MDV3100 PTM and MDV3100 | Day 1 through Day 72 (75 times)
  (Maximum concentration (observed))Cmax, (Area Under Curve from the time of dosing to the last measurable concentration)AUC0-t, (AUC extrapolated to infinity)AUC0-inf
Assessment of the pharmacokinetic profile of omeprazole (CYP2C19 substrate) in combination with MDV3100 PTM and MDV3100 | Day 1 through Day 72 (75 times)
  (Maximum concentration (observed))Cmax, (Area Under Curve from the time of dosing to the last measurable concentration)AUC0-t, (AUC extrapolated to infinity)AUC0-inf
Assessment of the pharmacokinetic profile of midazolam (CYP3A4 substrate) in combination with MDV3100 PTM and MDV3100 | Day 1 through Day 72 (75 times)
  (Maximum concentration (observed))Cmax, (Area Under Curve from the time of dosing to the last measurable concentration)AUC0-t, (AUC extrapolated to infinity)AUC0-inf

SECONDARY OUTCOMES:
Assessment of the pharmacokinetic profile of substrates pioglitazone (CYP2C8 substrate), S-warfarin (CYP2C9 substrate), omeprazole (CYP2C19 substrate), and midazolam (CYP3A4 substrate) in combination with MDV3100 PTM and MDV3100 | Day 1 through Day 72 (75 times)
  (Time to attain Cmax)tmax (Apparent terminal elimination half-life)t1/2, (Apparent total body clearance after extravascular dosing)CL/F, (Apparent volume of distribution during the terminal phase after extravascular dosing)Vz/F, Cmax, AUC0-t, AUC0-inf, (Pre-dose plasma concentration)C0h, (Minimum concentration (observed))Cmin, (AUC between two consecutive doses at steady-state)AUCtau, (Peak-trough ratio)PTR
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG) and clinical safety laboratory and, adverse events | Day 1 through Day 97

CONTACTS AND LOCATIONS:
Overall Officials: Operation Senior Research Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (2):
- South Africa (2):
  - Parexel, George
  - Parexel/Qdot Pharma, Port Elizabeth

REFERENCES:
- [Derived] Gibbons JA, de Vries M, Krauwinkel W, Ohtsu Y, Noukens J, van der Walt JS, Mol R, Mordenti J, Ouatas T. Pharmacokinetic Drug Interaction Studies with Enzalutamide. Clin Pharmacokinet. 2015 Oct;54(10):1057-69. doi: 10.1007/s40262-015-0283-1. PMID 25929560
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=22